CLINICAL TRIAL: NCT02078284
Title: Dose Escalation Study Evaluating the Safety of Dimethyl Sulfoxide Cryopreserved Platelets Compared With Liquid Stored Platelets in Patients With Uncontrolled Bleeding
Brief Title: Phase 1 Safety Study of Dimethyl Sulfoxide Cryopreserved Platelets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-12-04; CPP1-05 (Other: Army)
Record Dates: First submitted 2014-02-26; First posted 2014-03-05 (Estimated); Results first posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Thrombocytopenia
Keywords: platelet transfusion
MeSH Terms: conditions — Thrombocytopenia | interventions — 6-chloro-2-(1-piperazinyl)pyrazine; Dimethyl Sulfoxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Cohort 1 with 0.5 units of CPP (Experimental): A single 30 to 60 minute intravenous (IV) infusion of 0.5 unit of dimethyl sulfoxide (DMSO) cryopreserved platelets (CPP)
  Interventions: Biological: CPP
- Cohort 1 with 1 unit of LSP (Active Comparator): A single 30 to 60 minute intravenous (IV) infusion of 1 unit of liquid stored platelets (LSP)
  Interventions: Biological: LSP
- Cohort 2 with 1 unit of CPP (Experimental): A single 30 to 60 minute intravenous (IV) infusion of 1 unit of dimethyl sulfoxide (DMSO) cryopreserved platelets (CPP)
  Interventions: Biological: CPP
- Cohort 2 with 1 unit of LSP (Active Comparator): A single 30 to 60 minute intravenous (IV) infusion of 1 unit of liquid stored platelets (LSP)
  Interventions: Biological: LSP
- Cohort 3 with 2 units of CPP (Experimental): A single 30 to 60 minute intravenous (IV) infusion of 2 units of dimethyl sulfoxide (DMSO) cryopreserved platelets (CPP)
  Interventions: Biological: CPP
- Cohort 3 with 1 unit of LSP (Active Comparator): A single 30 to 60 minute intravenous (IV) infusion of 1 unit of liquid stored platelets (LSP)
  Interventions: Biological: LSP
- Cohort 4 with 3 units of CPP (Experimental): A single 30 to 60 minute intravenous (IV) infusion of 3 units of dimethyl sulfoxide (DMSO) cryopreserved platelets (CPP)
  Interventions: Biological: CPP
- Cohort 4 with 1 unit of LSP (Active Comparator): A single 30 to 60 minute intravenous (IV) infusion of 1 unit of liquid stored platelets (LSP
  Interventions: Biological: LSP

INTERVENTIONS:
Biological: CPP — One unit of frozen CPP contains approximately 3.4 x 10^11 irradiated platelets and approximately 6% DMSO in sterile 0.9% sodium chloride solution (total volume of 20 mL to 35 mL) stored frozen at ≤ -65°C.
  Other Names: dimethyl sulfoxide (DMSO) cryopreserved platelets (CPP)
  Arms: Cohort 1 with 0.5 units of CPP; Cohort 2 with 1 unit of CPP; Cohort 3 with 2 units of CPP; Cohort 4 with 3 units of CPP
Biological: LSP
  Other Names: liquid stored platelets (LSP)
  Arms: Cohort 1 with 1 unit of LSP; Cohort 2 with 1 unit of LSP; Cohort 3 with 1 unit of LSP; Cohort 4 with 1 unit of LSP

SUMMARY:
This study is to evaluate the safety of intravenous (IV) infusion of dimethyl sulfoxide (DMSO) cryopreserved platelets (CPP) in participants with World Health Organization (WHO) Grade 2 bleed in spite of receiving a transfusion of liquid stored platelets (LSP) in the past 48 hours by collecting adverse events (AEs) and by evaluating coagulation-related parameters to assess the evidence of any thrombotic events after CPP or LSP transfusion.

DETAILED DESCRIPTION:
After determining eligibility for study participation, 4 sequential cohorts of subjects will receive escalating doses of CPP (Test) or 1 unit of LSP (Control) randomized 6:1 within each cohort. Each sequential cohort will receive the following transfusions starting with the first cohort: 0.5, 1, 2, and 3 units of CPP with an additional single subject in each cohort who will receive 1 unit of LSP for a total of 28 subjects. Assignment to Test and Control platelets for subjects in each cohort will be centrally randomized using an interactive web response system (IWRS). Following the study transfusion, subjects are followed for evidence of transfusion reactions, thrombotic events, other AEs, coagulation-related parameters, and platelet efficacy endpoints. CPP or LSP will be transfused into a patient according to the randomized product and dose assignment within the cohort. Following the transfusion, subjects are followed for the remainder of Study Day 1 and on Study Day 2 for AEs and tested for coagulation markers including fibrinogen, D-dimer, prothrombin fragments 1 + 2 (F 1+2), thrombin antithrombin (TAT), anti-thrombin (AT), prothrombin time (PT), activated partial thromboplastin time (aPTT), thrombin generation testing (TGT) results, thromboelastography (TEG) results, and other potential complications of platelet transfusion such as transfusion reactions and thrombotic events including assessment of vital signs (blood pressure, heart rate, respiration rate, and pulse oximetry). A subject is considered to have completed the study for safety evaluation for dose escalation, if he/she receives a study infusion and completed study-related Day 3 procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age.
* Ability to comprehend the study procedures and signed informed consent.
* If pre-menopausal female, must have a negative serum pregnancy test, and, if of child bearing potential, must be using an acceptable method of contraception.
* Diagnosed with any the following: acute leukemia (ALL or AML), chronic leukemia (CML, CLL, CMML, or hairy cell leukemia), myelodysplasia, aplasia, hematopoietic or non-hematopoietic solid tumor, or therapy (chemotherapy or radiation) induced bone marrow aplasia or hypoplasia. Either autologous or allogeneic bone marrow transplant or peripheral or cord blood stem cell recipients may be enrolled.
* WHO grade 2 or greater bleeding.

Exclusion Criteria:

* Acute or chronic DIC as evidence by D-dimer greater than 8 μg/mL and fibrinogen less than 100 mg (0.1 g)/dL. Both criteria must be met. If data are in the medical record for fibrin degradation products (FDPs), then FDP must be <=40 μg/mL (FDP >40 μg/mL is indicative of DIC).
* PT or aPTT > 1.3 times the upper limit of normal for the laboratory.
* History of major operative procedures that required general anesthesia in the past 2 weeks.
* History of any prior major unprovoked thrombotic events and/or known inherited disorder of coagulation or platelet function (by history) (not to include clots in catheters, etc).
* A history or diagnosis of immune thrombocytopenia, thrombotic thrombocytopenic purpura, or hemolytic uremic syndrome.
* Females who are breastfeeding.
* Veno-occlusive disease or possible veno-occlusive disease.
* Receiving active, inpatient treatment with anti-platelet drugs and/or full anticoagulation therapy. Note: a heparin flush may be given daily and before and after blood draws to patients with a central line to keep the line patent.
* Subject previously enrolled in this study and received a study transfusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-11-05 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherrill J Slichter, MD, Principal Investigator — Bloodworks; Terry B Gernsheimer, MD, Principal Investigator — University of Washington, Division of Hematology; Zbigniew Szczepiorkowski, MD, PhD, Principal Investigator — Center for Transfusion Medicine Research, Lebanon, NH; Jose A Cancelas-Perez, MD, PhD, Principal Investigator — Hoxworth Blood Center
Locations (4):
- United States (4):
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hoxworth Blood Center, Cincinnati, Ohio
  - Puget Sound Blood Center, Seattle, Washington
  - University of Washington, Division of Hematology, Seattle, Washington

REFERENCES:
- [Derived] Slichter SJ, Dumont LJ, Cancelas JA, Jones M, Gernsheimer TB, Szczepiorkowski ZM, Dunbar NM, Prakash G, Medlin S, Rugg N, Kinne B, Macdonald VW, Housler G, Valiyaveettil M, Hmel P, Ransom JH. Safety and efficacy of cryopreserved platelets in bleeding patients with thrombocytopenia. Transfusion. 2018 Sep;58(9):2129-2138. doi: 10.1111/trf.14780. PMID 30204953

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who were admitted to the site's medical center and undergoing treatment for a hematologic malignancy were potentially eligible for the study. Potential study subjects were recruited by preliminary medical chart review against the study eligibility criteria.
Pre-assignment Details: Patient 29 was randomized to receive 0.5 Units of CPP but inadvertently received 1 Unit. This patient's data was analyzed with the 1 Unit CPP group.
Groups:
- 1 Unit of LSP: A single 30 to 60 minute intravenous (IV) infusion of 1 unit of liquid stored platelets (LSP)
Period: Overall Study
Arm/Group | Cohort 1 With 0.5 Units of CPP | Cohort 2 With 1 Unit of CPP | Cohort 3 With 2 Units of CPP | Cohort 4 With 3 Units of CPP | 1 Unit of LSP
Started | 5 | 7 | 6 | 6 | 4
Completed | 5 | 7 | 6 | 6 | 4
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patient 29 was randomized to receive 0.5 Units of CPP but inadvertently received 1 Unit. This patient's data was analyzed with the 1 Unit CPP group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 With 0.5 Units of CPP | Cohort 2 With 1 Unit of CPP | Cohort 3 With 2 Units of CPP | Cohort 4 With 3 Units of CPP | 1 Unit of LSP | Total
Number analyzed (Participants) | 5 | 7 | 6 | 6 | 4 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (17.3) | 57.7 (18.6) | 52.3 (15.8) | 53.3 (13.0) | 46.3 (16.2) | 51.9 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Patient 29 was randomized to receive 0.5 Units of CPP but inadvertently received 1 Unit. This patient's data was analyzed with the 1Unit CPP group.
  Participants
    Female | 4 | 2 | 3 | 1 | 1 | 11
    Male | 1 | 5 | 3 | 5 | 3 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 7 | 5 | 6 | 4 | 27
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 1 | 0 | 1 | 0 | 2
  White | 4 | 6 | 4 | 5 | 2 | 21
  More than one race | 1 | 0 | 0 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 7 | 6 | 6 | 4 | 28
Baseline Weight (kg) [Mean (Standard Deviation); unit: kg] | 91.4 (15.3) | 87.2 (23.9) | 87.7 (28.3) | 97.8 (16.4) | 81.1 (11.4) | 89.5 (20.1)
Baseline Height (cm) [Mean (Standard Deviation); unit: cm] | 171 (2.77) | 172 (8.55) | 176 (11.7) | 180 (11.6) | 177 (13.4) | 175.2 (10.0)

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events (AEs) by Level of Severity
Description: Clinical laboratory [chemistry (serum creatinine, lactate dehydrogenase (LDH), and troponin, and hematology (hemoglobin and hematocrit)] parameters, physical examination findings, electrocardiogram (ECG)] and vital sign AEs summarized by severity.
Time Frame: day of thru 6 days after transfusion
Population: as for baseline characteristics
Measure: Number; unit: adverse events
Arm/Group | Cohort 1 With 0.5 Units of CPP | Cohort 2 With 1 Unit of CPP | Cohort 3 With 2 Units of CPP | Cohort 4 With 3 Units of CPP | 1 Unit of LSP
Number analyzed (Participants) | 5 | 7 | 6 | 6 | 4
adverse events
  Total number of AEs | 8 | 18 | 6 | 21 | 5
  Total mild AEs | 6 | 11 | 1 | 9 | 5
  Total moderate AEs | 1 | 3 | 5 | 5 | 0
  Total Severe AEs | 0 | 1 | 0 | 1 | 0
  Total Life-threatening or Fatal AEs | 1 | 3 | 0 | 6 | 0

2. Primary Outcome: Number of Subject Who Experienced Adverse Events (AEs) for a Specific Severity
Description: Number of subjects who experienced AEs at specific levels of severity. Clinical laboratory [chemistry (serum creatinine, lactate dehydrogenase (LDH), and troponin, and hematology (hemoglobin and hematocrit)] parameters, physical examination findings, electrocardiogram (ECG)] and vital signs were evaluated.
Time Frame: day of thru 6 days after transfusion
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 With 0.5 Units of CPP | Cohort 2 With 1 Unit of CPP | Cohort 3 With 2 Units of CPP | Cohort 4 With 3 Units of CPP | 1 Unit of LSP
Number analyzed (Participants) | 5 | 7 | 6 | 6 | 4
Participants
  Total Patients with Any AE | 4 | 6 | 3 | 5 | 1
  Total Patients with any AE | 4 | 6 | 3 | 5 | 1
  Total Patients with Mild AEs | 4 | 4 | 1 | 5 | 1
  Total Patients with Moderate AEs | 1 | 1 | 3 | 1 | 0
  Total Patients with Severe AEss | 0 | 1 | 0 | 1 | 0
  Total Patients with Life-threatening or Fatal AEs | 1 | 1 | 2 | 2 | 0
  Related to Investigational Product | 1 | 2 | 2 | 2 | 0

3. Primary Outcome: Number of Subject With Thrombotic Events
Description: Subjects with any signs or symptoms of thrombotic events.
Time Frame: 6 days after transfusion
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 With 0.5 Units of CPP | Cohort 2 With 1 Unit of CPP | Cohort 3 With 2 Units of CPP | Cohort 4 With 3 Units of CPP | 1 Unit of LSP
Number analyzed (Participants) | 5 | 7 | 6 | 6 | 4
Participants | 0 | 0 | 0 | 0 | 0

4. Other Pre Specified Outcome: Corrected Count Increments (CCI)
Description: Corrected Count Increments Expressed in units of mm^2/(µL*10¹¹ platelets) (CCI) in the 6 hour period after the study platelet transfusion and on Day 2 (approximately 24 hours after the study platelet transfusion)
Time Frame: Day 1 up to 6 hrs after transfusion and Day 2 approx 24 hrs after transfusion
Measure: Mean (Standard Deviation); unit: mm^2/(μL*1011 platelets)
Arm/Group | Cohort 1 With 0.5 Units of CPP | Cohort 2 With 1 Unit of CPP | Cohort 3 With 2 Units of CPP | Cohort 4 With 3 Units of CPP | 1 Unit of LSP
Number analyzed (Participants) | 5 | 7 | 6 | 6 | 4
mm^2/(μL*1011 platelets)
  CII: Day 1 up to 6 hrs after | 2.40 (5.76) | 3.10 (2.92) | 2.73 (1.51) | 3.70 (2.34) | 14.8 (9.66)
  CII: Day 2 | 5.19 (6.22) | -2.05 (4.96) | 5.63 (7.05) | 2.35 (3.94) | 4.13 (3.58)

5. Other Pre Specified Outcome: Count Increment
Description: Count Increment expressed in units of platelets (x10^3 µL) (CI)
Time Frame: On Day 1 up to 6 hours after transfusion and on Day 2 approximately 24 hours after transfusion
Measure: Mean (Standard Deviation); unit: platelets*10^3 µL
Arm/Group | Cohort 1 With 0.5 Units of CPP | Cohort 2 With 1 Unit of CPP | Cohort 3 With 2 Units of CPP | Cohort 4 With 3 Units of CPP | 1 Unit of LSP
Number analyzed (Participants) | 5 | 7 | 6 | 6 | 4
platelets*10^3 µL
  Day 1 Up to 6 Hours After | 1.20 (3.11) | 3.67 (2.42) | 6.50 (3.89) | 13.2 (6.38) | 30.5 (20.3)
  Day 2 | 2.80 (3.11) | -2.57 (6.40) | 12.5 (14.2) | 10.7 (13.3) | 8.75 (7.97)

ADVERSE EVENTS:
Time Frame: Day of transfusion thru 6 days after transfusion
Arm/Group | Cohort 1 With 0.5 Units of CPP | Cohort 2 With 1 Unit of CPP | Cohort 3 With 2 Units of CPP | Cohort 4 With 3 Units of CPP | 1 Unit of LSP
All-Cause Mortality (participants affected / at risk) | 1/5 | 1/7 | 0/6 | 1/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/5 | 2/7 | 0/6 | 2/6 | 0/4
Other Adverse Events (participants affected / at risk) | 4/5 | 6/7 | 3/6 | 5/6 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 With 0.5 Units of CPP (N=5) | Cohort 2 With 1 Unit of CPP (N=7) | Cohort 3 With 2 Units of CPP (N=6) | Cohort 4 With 3 Units of CPP (N=6) | 1 Unit of LSP (N=4)
Adults respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prolonged QT interval (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis with gram negative rod bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Worsening lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Worsening sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 With 0.5 Units of CPP (N=5) | Cohort 2 With 1 Unit of CPP (N=7) | Cohort 3 With 2 Units of CPP (N=6) | Cohort 4 With 3 Units of CPP (N=6) | 1 Unit of LSP (N=4)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Affect lability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Belligerence (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electocardiogram abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Respiratory rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scrotal eodema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin odor abnormal (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Unresponsive to stimuli (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No